CLINICAL TRIAL: NCT00649220
Title: Prospective, Single-arm, Multi-centre, Open-label Study to Investigate the Potential to Reduce Concomitant Antipsychotics Use in Patients With Moderate to Severe Dementia of Alzheimer's Type (DAT) Treated With Memantine
Brief Title: Memantine and Antipsychotics Use
Acronym: MemAP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to too slow enrollment
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRZ 90001-0716/1; 2007-004489-41 (EudraCT Number)
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Results first posted 2011-09-13 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Memantine (Experimental)
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — memantine tablets, twice a day (bid), for 20 weeks

SUMMARY:
To investigate the potential to reduce concomitant antipsychotic medication use in subjects with moderate dementia of Alzheimer's type, treated with memantine.

ELIGIBILITY:
Inclusion criteria:

* Current diagnosis of probable Alzheimer's disease consistent with NINCDS-ADRDA criteria or with DSM IV TR criteria for Dementia of the Alzheimer's type.
* MRI or CT scan supporting the diagnosis of DAT without indications of any relevant other CNS disorders.
* Patients treated with any acetylcholinesterase inhibitor (AChEI) man be included.
* The patient should have German as a mother-tongue or at least speak the language fluently.

Exclusion criteria:

* Evidence (including CT/MRI results) of any clinically significant central nervous system disease other than Alzheimer's disease.
* Modified Hachinski Ischemia score greater than 4 at screening.
* Intake of any medication that is contra-indicated in combination with memantine.
* Treatment with depot antipsychotics.
* History of severe drug allergy, or hypersensitivity, or patients with known hypersensitivity to memantine, amantadine or lactose.
* Known or suspected history of alcoholism or drug abuse within the past 10 years.
* Previous treatment with memantine or participation in an investigational study with memantine.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-07; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (1):
- Alexianer Hospital, Krefeld, North Rhine-Westphalia, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Memantine: Memantine tablets, twice a day (bid).
Period: Overall Study
Arm/Group | Memantine
Started | 19
Completed | 16
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Memantine
Number analyzed (Participants) | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 72.4 (9.7)
Age, Customized [Number; unit: participants]
  Between 50 and 85 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Region of Enrollment [Number; unit: participants]
  Germany | 19

OUTCOME MEASURES:

1. Primary Outcome: Maximum Dose Reduction of Antipsychotics (AP) in Percent of Defined Daily Dose (DDD) From Baseline to a Post-baseline Visit at Which the Value of the Visual Analogue Scale (VAS) Compared With the Baseline Value Was =< 15 Percent.
Description: VAS: see #8. Mean "percent of the total Defined Daily Dose (DDD)", averaged over one week, was calculated. Total DDD was calculated as sum of DDD for each AP drug. DDD is the assumed average maintenance dose per day defined by WHO. The reduction of AP Δ [percent] was calculated as a difference between the mean total DDD recorded at baseline and the mean total DDD recorded at the respective week. Measurements from those post-baseline visits were taken into account only when the value of the VAS was not substantially worse compared to baseline.
Time Frame: Week 8-20 post baseline
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Percent of daily dose [DDD]
Arm/Group | Memantine
Number analyzed (Participants) | 19
Percent of daily dose [DDD] | -13.9 (13.58) [-20.4 to -7.36]
Statistical Analysis 1: Comparison: Memantine; Two-side, paired t-test on the null hypothesis that antipsychotics are reduced by 10% compared to baseline; Test type: Superiority or Other; p = 0.22626, t-test, 2 sided
Statistical Analysis 2: Comparison: Memantine; Wilcoxon signed rank test on the null hypothesis that antipsychotics are reduced by 10% compared to baseline; Test type: Superiority or Other; p = 0.34192, Wilcoxon signed rank test

2. Secondary Outcome: Reduction of Antipsychotic Drug Dose From Baseline to Week 8, 12, 16 and/or 20.
Description: See #1 and #8. Change of <0 reveals a reduction of AP compared to baseline.
Time Frame: Week 8-20 post Baseline
Population: Intention to treat (ITT).
  Week 8: n=16; Week 12: n=14; Week 16: n=13; Week 20: n=15
Measure: Mean (Standard Deviation); unit: Percent of daily dose [DDD]
Arm/Group | Memantine
Number analyzed (Participants) | 15
Percent of daily dose [DDD]
  Week 8 | -4.4 (5.53)
  Week 12 | -8.2 (12.38)
  Week 16 | -10.6 (13.49)
  Week 20 | -14.9 (15.05)

3. Secondary Outcome: Change in the Mini-Mental State Examination (MMSE) Score Value From Baseline to Week 20.
Description: MMSE is a brief, physician-administered scale, designed for measuring the cognitive functions, such as: orientation, memory, attention, naming, and comprehension. The scoring range of MMSE is 0 to 30 points. A score of 23 or lower is indicative of cognitive impairment. Change of >0 reveals an improvement compared to baseline.
Time Frame: Week 20 post baseline
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 15
units on a scale | 0.9 (3.44) [-1.04 to 2.77]

4. Secondary Outcome: Change of "Test for the Early Detection of Dementia With Discrimination From Depression [TE4D]" Score Value From Baseline to Week 4, 8, 12, 16, and/or 20 - First Part: Total Dementia
Description: TE4D is a psychometric, physician-administered test that is used for both screening subjects with early dementia and monitoring the clinical progress of the disease. The first part consists of 9 items, which assess different symptoms associated with dementia such as memory, time-orientation, etc. The scoring range is 0 to 50 points. A score of 35 or lower is an indication of dementia.
  A change >0 represents an improvement.
Time Frame: Week 4-20 post baseline
Population: Intent to treat (ITT).
  Week 4: n=18; Week 8: n=17; Week 12: n=16; Week 16: n=16; Week 20: n=17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 17
units on a scale
  Week 4 | -2.3 (7.64)
  Week 8 | -0.3 (5.31)
  Week 12 | -1.3 (4.48)
  Week 16 | 0.7 (5.39)
  Week 20 | 1.4 (4.2)

5. Secondary Outcome: Change of "Test for the Early Detection of Dementia With Discrimination From Depression [TE4D]" Score Value From Baseline to Week 4, 8, 12, 16, and/or 20 - Second Part: Total Depression
Description: TE4D is a psychometric, physician-administered test that is used for both screening subjects with early dementia and monitoring the clinical progress of the disease. The second part consists of a proxy rating and a self-assessment rating. The scoring range of each rating is 1 to 10. The maximum total score of 10 corresponds to severe depression.
  A change <0 reveals an improvement compared to baseline.
Time Frame: Week 4-20 post Baseline
Population: Intention to treat (ITT).
  Week 4: n=18; Week 8: n=17; Week 12: n=16; Week 16: n=16; Week 20: n=17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 17
units on a scale
  Week 4 | 2.5 (4.84)
  Week 8 | 1.6 (3.97)
  Week 12 | -0.1 (3.26)
  Week 16 | -0.2 (2.07)
  Week 20 | -0.4 (2.09)

6. Secondary Outcome: Change of Modified Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADLB19) Score Value From Baseline to Week 4, 8, 12, 16, and/or 20.
Description: The modified ADCS-ADL19 is comprehensive battery of ADL questions aimed to measure the functional ability of subjects with Dementia of Alzheimer's type over a broad range of dementia severity. It has a scoring range of 0 to 54 with the lower scores indicating greater functional impairment. Each ADL item was rated from the highest level of independent performance to complete loss.
  Change of >0 reveals an improvement compared to baseline.
Time Frame: Week 4-20 post Baseline
Population: Intention to treat (ITT).
  Week 4: n=18; Week 8: n=17; Week 12: n=16; Week 16: n=16; Week 20: n=18
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Memantine
Number analyzed (Participants) | 18
Units on a Scale
  Week 4 | -0.7 (6.33)
  Week 8 | 2.2 (8.09)
  Week 12 | 3.8 (11.07)
  Week 16 | 3.8 (11.27)
  Week 20 | 2.4 (11.08)

7. Secondary Outcome: Change of Nurses' Observation Scale for Geriatric Patients [NOSGER] Total Score Value From Baseline to Week 4, 8, 12, 16, and/or 20
Description: NOSGER is a comprehensive scale, which contains 30 items of behavior, each rated on a 5-point scale according to the frequency of occurrence by direct observation. Item scores are summarized into 6 dimension scores: memory, instrumental activities of daily life, self-care, mood, social behavior, and disturbing behavior. The NOSGER has a scoring range of 30 to 150 with the higher scores indicating worse subject's status. The items in each group are rated for their frequency ranging from 1 (never) to 5 (always).
  A change of <0 reveals an improvement compared to baseline.
Time Frame: Week 4-20 post Baseline
Population: Intention to treat (ITT).
  Week 4: n=18; Week 8: n=17; Week 12: n=16; Week 16: n=16; Week 20: n=17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 18
Units on a scale
  Week 4 | -0.4 (10.9)
  Week 8 | -2.1 (10.31)
  Week 12 | -5.4 (13.29)
  Week 16 | -8.4 (18.74)
  Week 20 | -7.9 (19.02)

8. Secondary Outcome: Change in the VAS Score From Baseline to Week 8, 12, 16 and/or 20.
Description: VAS is a report device to measure the subject's burden caused by behavioral symptoms. To measure the burden on the VAS only the first 3 items of the Neuropsychiatric Inventory (NPI) Questionnaire were considered (delusions, hallucinations (visual and auditory), and agitation / aggression). The VAS consists of a 100 mm horizontal line, anchored at the ends with the reference "not at all" and "extremely". The VAS score was determined by measuring in mm from the left hand end of the line to the point, where the investigator had marked the magnitude of a subject's burden.
Time Frame: Week 8-20 post Baseline
Population: Intention to treat (ITT).
  Week 8: n=17; Week 12: n=16; Week 16: n=16; Week 20: n=18
Measure: Mean (Standard Deviation); unit: Units on a scale [cm]
Arm/Group | Memantine
Number analyzed (Participants) | 18
Units on a scale [cm]
  Week 8 | -1.5 (1.94)
  Week 12 | -1.7 (2.53)
  Week 16 | -1.2 (2.86)
  Week 20 | -1.4 (2.46)

ADVERSE EVENTS:
Time Frame: All SAEs/AEs from baseline until 4 weeks after end of treatment (in total 20 weeks)
Description: The table of "Other Adverse Events" includes all non-serious AEs. The investigator asked the patient for AEs systematically at each visit.
Arm/Group | Memantine
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=19)
Depression (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Sleep Disturbances (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=19)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Listless (Psychiatric disorders) | 1 (1)
Sleep-related eating disorder (Psychiatric disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to too slow enrollment lead to a small sample size, limiting the ability for confirmatory analysis. All analysis of the primary efficacy endpoint were treated as exploratory.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No results to be published without written agreement by sponsor; manuscripts to be sent to sponsor at least 6 weeks before submission. Sponsor to give written opinion within 30 days. Sponsor is entitled to exert influence on the contents of publications, to postpone publications up to 36 months after end of the study, and to name co-authors. In case of justified doubts of sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.